CLINICAL TRIAL: NCT00320827
Title: Phase 1 Study of CS-1008, a Humanized Monoclonal Antibody Targeting Death Receptor 5 (DR5), Administered Weekly to Patients With Advanced Solid Malignancies and Lymphomas (Without Leukemic Component)
Brief Title: Study of CS-1008 in Patients With Advanced Solid Malignancies and Lymphomas (Without Leukemic Component)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1008-A-U101
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Malignancies; Lymphoma
Keywords: Apoptosis; Death receptor 5; Cancer; Advanced solid malignancies and lymphomas (without leukemic component)
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — tigatuzumab

INTERVENTIONS:
Drug: CS-1008 (humanized anti-DR5 antibody)

SUMMARY:
This is a dose escalation study of CS-1008 (humanized anti-DR5 antibody) to determine the recommended Phase 2 dose and the maximum tolerated dose. Drug will be administered for six weeks and possibly up to 12 weeks depending on response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed metastatic solid tumors or lymphomas (with no leukemic component) which are refractory to, not curable with, or not eligible for standard treatment(s).
* Eighteen years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status equal to or less than 2
* Resolution of any toxic effects (except alopecia) of prior therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 grade of equal to or less than 1
* Men and women of childbearing potential must be willing to consent to use effective contraception while on treatment and for at least 3 months thereafter.
* All female patients of childbearing potential must have a negative pregnancy test (serum or urine) within 3 days prior to treatment
* Patients must be fully informed about their illness and the investigational nature of the study protocol

Exclusion Criteria:

* Anticipation of the need for a major surgical procedure or radiation therapy during the study
* Treatment with chemotherapy, hormonal therapy, radiotherapy, major surgery, or any investigational agent within 4 weeks (6 weeks for nitrosoureas, mitomycin C, immunotherapy, biological therapy, or major surgery) of study enrollment
* Cumulative radiation therapy to greater than 25% of the total bone marrow
* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other clinically significant thromboembolytic event; clinically significant pulmonary disease (e.g., severe chronic obstructive pulmonary disease [COPD] or asthma)
* Patients with a clinically active brain metastasis (i.e., not treated or still requiring therapy with steroids or radiotherapy [RT]; or with progression 4 weeks after the completion of RT) or an uncontrolled seizure disorder, spinal cord compression, or carcinomatous meningitis
* Clinically significant active infection which requires antibiotic therapy, or HIV-positive patients receiving antiretroviral therapy.
* Chronic diarrhea, inflammatory bowel disease, or partial bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
To determine the recommended Phase 2 dose

SECONDARY OUTCOMES:
To investigate the pharmacokinetics of CS-1008 administered weekly
To characterize the immunogenicity of CS-1008 by monitoring for anti-CS-1008 antibodies
To study potential biomarkers of CS-1008 activity
To make preliminary assessments of anti-tumor effects of CS-1008

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States